CLINICAL TRIAL: NCT07404566
Title: The Merits of Implementing microRNAs for Diagnosing Hepatocellular Carcinoma Among Hepatitis C Patients
Brief Title: Utility of MicroRNAs for Diagnosing Hepatocellular Carcinoma in Hepatitis C Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Raafat R. Mohammed, Assistant consultant of Clinical Pathology, Benha University
Other Study IDs: E/C.S/N.R15/2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The study involved the collection of human blood samples, specifically processed into the following formats:
  Serum: Obtained by collecting blood in clean tubes, allowing it to clot, and centrifuging at 1000 rpm for 10 minutes.
  Plasma/Supernatant: Collected into EDTA-containing tubes and centrifuged to separate the supernatant.
  Total RNA: Extracted from the blood samples, specifically including the microRNA fraction for PCR analysis.
  Storage and Laboratory Processing
  Serum Storage: Serum samples used for alpha-fetoprotein (AFP) ELISA estimation were kept frozen at -20 °C.
  RNA Storage: The supernatant for RNA extraction was stored in RNase-free tubes at -80 °C prior to the extraction process.
  Molecular Analysis: The retained specimens were used for reverse transcription of cDNA and subsequent Real-time RT-qPCR to determine the relative number of Mir copies using the ΔΔCT method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCV Group: 21 patients with newly diagnosed or chronic HCV infection, free of findings suggestive of cirrhosis or HCC.
  Interventions: Diagnostic Test: PCR
- LC Group: 21 patients with HCV complicated by liver cirrhosis.
  Interventions: Diagnostic Test: PCR
- HCC Group: 21 patients with HCV complicated by hepatocellular carcinoma.
  Interventions: Diagnostic Test: PCR
- Control Group: 21 healthy volunteers who passed pre-donation investigations at a Blood Bank.
  Interventions: Diagnostic Test: PCR

INTERVENTIONS:
Diagnostic Test: PCR — PCR quantification of plasma microRNA levels (MiR-21, 1246, 205, 29a-3p, and 497).

SUMMARY:
This study evaluates a target population of patients with Hepatitis C virus (HCV) infection, including those with complications like liver cirrhosis (LC) and hepatocellular carcinoma (HCC), to investigate the diagnostic utility of a specific panel of microRNAs (miRNAs). The intervention involves quantifying the plasma expression (PE) levels of MiR-21, 1246, 205, 29a-3p, and 497 via PCR and comparing them to healthy controls to determine their efficacy as biomarkers. The primary outcome is to assess the sensitivity, specificity, and overall accuracy of these miRNAs in differentiating HCC from cirrhotic and non-cirrhotic HCV cases, aiming to establish more reliable screening tools than current standard biomarkers like alpha-fetoprotein (AFP).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed HCV infection.
* Chronic uncomplicated HCV infection.
* HCV complicated with liver cirrhosis.
* HCV complicated with HCC on top of cirrhosis.
* Willingness to participate and sign written informed consent.

Exclusion Criteria:

* Advanced stage of hepatic cirrhosis with portal hypertension or hepatorenal failure.
* Hepatic malignancies other than HCC.
* Bilharzial pre-portal fibrosis.
* Alcoholic fatty liver disease
* hepatosteatosis.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals attending outpatient clinics for new or chronic HCV follow-up, and healthy volunteers from blood banks, primarily located in Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Success Rate of Diagnostic Regimens in Identifying Hepatocellular Carcinoma | Around 3 months
  iagnostic utility (sensitivity, specificity, and accuracy rate) of estimated plasma expression (PE) levels of microRNAs (specifically Mir-1246, Mir-21, and Mir-497) to distinguish HCC from LC and HCV

SECONDARY OUTCOMES:
Diagnostic Performance for LC | Around 3 months
  Differentiating liver cirrhosis using downregulated MiR-205 and overexpressed MiR-29a.
Biomarker Correlation | Around 3 months
  Correlation between miRNA levels and serum Alpha-Fetoprotein (AFP).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of medicine, Alexandria, El Alexandria, Egypt